CLINICAL TRIAL: NCT00167492
Title: Enteric Coated Mycophenolic Acid (Myfortic) in Liver Transplant Recipients- Effect on Compliance and Calcineurin Inhibitor and Corticosteroid Sparing
Brief Title: Enteric Coated Myfortic for Liver Transplant Recipients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Novartis (Industry)
Responsible Party: Dr. Bob Saggi, Memorial Hermann Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-05-0197; Novartis Pharmaceuticals; CERL080A-US11
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Myfortic — 720 mg by mouth every 12 hours

SUMMARY:
The purpose of this study is to replace the mycophenolate mofetil (Cellcept) which is our usual therapy after liver transplantation with sodium mycophenolic acid (Myfortic®) and to find out the effect this change may have on the development of side effects such as relief of gastrointestinal (stomach) problems. In the past we have had to stop Cellcept (our current drug) because of these side effects. We will also try to see if improved usage of this drug (Myfortic®) will allow us to use lower doses of other medications that lower your immune system. We will do some special tests on your blood to see if the amount of the drug is related with its effect on the immune system and side effects. Both Cellcept and Myfortic® are FDA approved medications although Myfortic® is not approved for use after liver transplantation. Myfortic® is really the same active drug as Cellcept® (Mycophenolic acid) but has been coated to prevent breakdown of the drug in the stomach and is made to lower the known gastrointestinal effects of Cellcept such as diarrhea, abdominal pain and nausea.

DETAILED DESCRIPTION:
Mycophenolic Acid (MPA) has been shown to be an effective immune suppressant in organ transplantation. Its gastrointestinal side effects, however, have limited its use in liver transplantation (OLT). A new form of MPA that is enteric coated (Myfortic) has been developed to address the issue of GI side effects. While considerable experience has been gained with this new formulation in kidney transplants (ref) the information regarding the use of Myfortic in OLT recipients is limited. The purpose of the study is to assess the safety and efficacy of Myfortic in OLT recipients. The study will include a close follow-up of the patients with regard to side effects and potential adverse effects of the drug. It will also monitor the rate of compliance with this medication among the patients in the study. The efficacy of the drug will be determined by the rate of rejection but also and more importantly by our ability to withdraw corticosteroids and minimize calcineurin inhibitors (CNI).

Several tests will be conducted as part of the study. Some of those are "Standard of Care" tests such as liver function tests and complete blood cell count (CBC). Some tests however, will be performed specifically for this study. These include a patient questionnaire to be filled at various time points and blood tests designed to assess the integrity of the immune system.

The benefit to the patients is three-fold:

The patients will receive the medication free of charge for the duration of the study.

The proven efficacy of MPA as an immune suppressant may allow us to reduce or eliminate the use of corticosteroids and/or CNI whose long and short-term side effects are major causes of morbidity in OLT recipients.

Avoidance of the GI side effects of non-enteric coated MPA, which is our standard drug in OLT.

The risks for the patient include the potential deleterious side effects of MPA, namely bone marrow depression, GI side-effects (nausea, diarrhea, abdominal pain), and infections.

The general benefits from the study may be the addition of a better formulation of MPA to the list of drugs used for immunosuppression in OLT. Additionally, routine use of this drug may minimize the long-term adverse effects of CNI and corticosteroids thus improving long-term patient survival and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients
* Age: 18-70
* Capable of oral intake

Exclusion Criteria:

* Hepatitis C Cirrhosis
* Hepatocellular Carcinoma T3
* Liver retransplantation
* Pregnancy
* Platelet count <40,000
* White Blood Cell count (WBC) <3,000
* Incapable of oral intake
* More than 30 days post op

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Rate of rejection | 6 months
Rate of gastrointestinal side-effects | 6 months

SECONDARY OUTCOMES:
Levels of calcineurin inhibitors | 6 months
Renal function | 6 months
Relationship of dose to biologic monitoring of immunosuppression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bob Saggi, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States